CLINICAL TRIAL: NCT06878287
Title: Bright Light Therapy During Residential Alcohol Withdrawal : a Double Blind Randomized Placebo Controlled Study
Brief Title: Bright Light Therapy During Residential Alcohol Withdrawal
Acronym: LUNA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D20-P49
Record Dates: First submitted 2024-09-27; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Light therapy every morning (8 am-8.30 am)
  Interventions: Other: Light exposure
- Control group (Placebo Comparator): Dim-Light exposure every morning (8 am-8.30 am)
  Interventions: Other: Placebo light

INTERVENTIONS:
Other: Light exposure — 30 minutes morning exposure to light (10 000 lux) using a light-box device filtering UV (CE marking)
  Arms: Experimental group
Other: Placebo light — 30 minutes exposure to the same device using a filter inactivating light intensity (< 10 lux)
  Arms: Control group

SUMMARY:
This is a randomized controlled trial assessing the effectiveness of light therapy versus placebo in patients undergoing alcohol withdrawal.

DETAILED DESCRIPTION:
All eligible patients will be offered and explained the study by a psychiatrist/addictologist during the consultation (or teleconsultation) to schedule a 14-day hospitalization for alcohol withdrawal (maximum 3 months before hospitalization). Patients will be randomized centrally to one of the following two treatment conditions (blind maintained by a nurse independent of the assessment), on day D0 of inpatient treatment for withdrawal (standardized withdrawal over 14 days with hydration, vitamin B1, benzodiazepines in gradual decrease before stopping and according to signs of withdrawal):

1. Active light therapy (10,000 Lux).
2. Placebo light therapy (with filter <10 Lux). Every morning in the room (patient in a single room), at 8 am, for 30 min, for the entire duration of withdrawal, i.e. 13 days (start on D1) and stopped on D14.

No change in usual care apart from this intervention.

After checking the inclusion and non-inclusion criteria and obtaining consent, patients will be randomized (ratio 1:1) between the groups with active light therapy or placebo, by connecting to a randomization website (REDCap software) using a randomization list prepared in advance, balanced by block of randomly variable size

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged from 18 to 65 years old and have a diagnosis of Alcohol Use Disorder
* Patients must be intreated for alcohol withdrawal, for at least two weeks
* Patients must report heavy drinking episodes in the past month
* Patients must be able to understand medical information and consent to the treatment
* Patients must be considering a goal of abstinence from alcohol

Exclusion Criteria:

* Ophthalmic pathology (cataract, macular degeneration, glaucoma, retinitis pigmentosa) and diseases affecting the retina (retinopathy, diabetes, herpes, etc.)
* Subjects who have already received light therapy in the last 6 months
* Lactating of pregnant women
* Psychiatric comorbidity requiring an intreatment, or risk of manic episode (subjects with depressive or anxious symptoms compatible with an out-treatment can be included)
* Substance Use Disorder other than alcohol and/or tobacco
* Severe cognitive impairment (MOCA < 10)
* Patients being under legal protection measure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol relapse or lapse | 4 and 12 weeks
  Assessment of alcohol intake at the follow-up visits using a Timeline Followback.
  Relapse : any heavy drinking day, i.e. 5 or more drinks/day for a man or 4 or more drinks/day for a woman, as defined by the NIAAA (2005) and the FDA (2015), and/or 14 drinks or more per week for at least 4 weeks.
  Lapse : any alcohol intake not meeting the criteria for relapse

SECONDARY OUTCOMES:
Actigraphy | 1 day and third week
  Wristwatch actigraph delivered at inclusion, which allows measurement of activity and sleep-wake parameters using an accelerometer worn on the wrist MotionWatch8 from CamNTech®
Alcohol withdrawal severity | 2 weeks
  Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-Ar) : maximum and mean score on the first 5 days after admission
Circadian typology | At inclusion
  Chronotype questionnaire (Horne & Östberg) a
Alcohol craving | At inclusion, 1, 2, 4 and 12 weeks
  Obsessive Compulsive Drinking Scale (OCDS)
Depressive and anxious symptomatology | At inclusion, 1, 2, 4 and 12 weeks
  * Montgomery-Åsberg Depression Rating Scale (MADRS)
  * Self-questionnaire : QIDS-SD16 and GAD-7
Suicidal risk | At inclusion, 1, 2, 4 and 12 weeks
  Columbia-Suicide Severity Rating Scale (C-SSRS)
Cognitive impairment | At inclusion, 2 and 12 weeks
  Montreal Cognitive Assessment (MoCA) : three different versions
Light therapy tolerance | At 2 weeks
  Side effects questionnaire designed for a previous study
Polysomnography | 1 week
  Sleep recording at the sleep laboratory, measuring :
  * Sleep stages
  * Total Sleep Time
  * Sleep Efficiency
  * Number of awakenings or arousals
  * Snoring
  * Apnea-Hypopnea Index (AHI)
  * Periodic Limb Movements
Subjective quality of sleep | 12 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Number of days with 2 drinks or more | 4, 12 weeks
  % of days with 2 drinks or more at the follow-up visits
Heavy drinking days | 4, 12 weeks
  % of heavy drinking days at the follow-up visits
Days with no drinking | 4, 12 weeks
  % of days with no drinking at the follow-up visits
Percent with complete abstinence | 4 and 12 weeks
  % of subjects with no drinking at the follow-up visits
Number of individuals in relapse | 4 , 12 weeks
  % of subjects meeting criteria for relapse at the follow-up visits
Sleep diary | From inclusion to third week
  sleep diary.give at the first appointment then fill in every day
Circadian typology | one day
  seasonal profile (SPAQ)
Actigraphy | one day to third week
  Wristwatch actigraph delivered at inclusion, which allows measurement of activity and sleep-wake parameters using an accelerometer worn on the wrist ScanWatch from Withings®
Alcohol withdrawal severity | one day to 2 weeks
  mean benzodiazepine dosage required by day during the 2 weeks of treatment
Subjective quality of sleep | one day, 2 day to12 weeks
  Insomnia Severity Index (ISI)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alexis GEOFFROY, PhD, Principal Investigator — University Hospital Group for Psychiatry and Neurosciences
Locations (1):
- Adult Emergency Department - Bichât Hospital, Paris, Île-de-France Region, France